CLINICAL TRIAL: NCT00228631
Title: Analysis of T-Cell Immune Reconstitution Following Allogeneic Hematopoietic Stem Cell Transplantation for Severe Sickle Cell Disease (ImmuneReconstSCD)
Brief Title: Analysis of T-Cell Immune Reconstitution Following Allogeneic Hematopoietic BMT for Severe SCD
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Ann E. Haight, Assistant Professor, Emory University
Other Study IDs: IRB00021821; 21821 (formerly 849-2005) (Other: Other)
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Sickle Cell Disease
Keywords: sickle; cell
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Sickle Cell Disease Bone Marrow Transplant: Sickle Cell Disease Bone Marrow Transplant candidates

SUMMARY:
In this study, patient blood samples from NMA transplants will be provided by Pittsburgh, and samples from myeloablative transplants will be provided by Atlanta (comparative controls). Samples would be obtained pre- and post-BMT from the recipient at a total of 7 timepoints, and from the donor at one timepoint.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is a serious inherited disorder of red blood cells that shortens life and causes life-long problems. One of the most common genetic diseases in America, SCD affects 1 of every 375 African-American live births, and can be identified by routine newborn screening. SCD manifests with vaso-occlusive events, the most common of which is the "sickle pain crisis," which causes severe and unrelenting pain, typically in the back, chest, or long bones. Other types of vaso-occlusive events involve the spleen, brain (stoke), retina, bones, kidney and lungs. Patients are at increased risk for death due to bacterial infections, damage to vital organs, or aplastic crisis (failure to produce any red cells), and often suffer chronic organ damage.

Patients with frequent and severe complications in early childhood are typically felt to be at highest risk for continued debilitating problems and early death. These severely affected children have been the subject of efforts to cure SCD through bone marrow transplantation (BMT) from a healthy donor. BMT is curative for SCD because it provides a source of normal hemoglobin production. BMT is performed by giving the patient high doses of chemotherapy, then infusing bone marrow from a healthy donor into a large vein in the recipient, followed by an intensive period of supportive care and immune suppression. Over 200 patients with SCD have been transplanted world-wide, primarily from sibling donors who are HLA (tissue or transplantation type) matched. Of those transplanted in a North American cooperative study, about 95% of these patients survived the transplant, and about 85% are free of sickle cell disease. The Atlanta program was the largest contributor to this study. Through 2004, Atlanta has transplanted 18 children with SCD from matched siblings; all are free of sickle cell disease and none have died.

Because conventional (myeloablative) BMT carries significant risks of morbidity and mortality ant thus limits its use, researchers have recently been investigating less risky methods of BMT for SCD, called reduced intensity or non-myeloablative (NMA) transplant. Dr. Catherine Wu of the Dana Farber Cancer Institute and Dr. Laksmannan Krishnamurti of the Children's Hospital of Pittsburgh are both performing NMA transplant for adults (Wu) and children (Krishnamurti) with severe SCD. In Atlanta (Haight), patients continue to be offered transplant using the conventional myeloablative approach.

Important questions remain about the functional and long-term status of transplanted SCD patients in a variety of areas; this study will focus upon immune function. Because little is know about the functional immune status of patients after non-myeloablative transplants, and certainly not those who undergo transplantation for the diagnosis of sickle cell anemia, patient blood samples will be analyzed for extent of immune reconstitution following transplant through immunophenotyping of various immune cell subsets, molecular analysis of reconstitution of T cell neogenesis (TREC analysis) and T cell receptor complexity (TCR Vbeta spectratyping).

ELIGIBILITY:
Inclusion Criteria:

Undergoing allogeneic bone marrow transplantation for sickle cell disease.

Exclusion Criteria:

-

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: At in-patient or out-patient transplant clinic (All sickle cell disease bone marrow transplant patients will be offered participation)
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2005-09; Primary Completion 2011-08 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
To determine the rate of T cell immune reconstitution in children with sickle cell disease | 1 year after accrual closed

CONTACTS AND LOCATIONS:
Overall Officials: Ann Haight, MD, Principal Investigator — Children's Healthcare of Atlanta/Emory
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States